CLINICAL TRIAL: NCT00044460
Title: A 24-week Randomized, Double-Blind, Parallel-Group, Multicenter Study to Demonstrate the Efficacy and Safety of Two Different Rosiglitazone Dosing Regimens, 4mg OD and 8mg OD, in Poorly-Controlled Drug Naive Patients With Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety In Poorly Controlled Type 2 Diabetics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 49653/326
Record Dates: First submitted 2002-08-29; First posted 2002-08-30 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes drug-naive
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rosiglitazone

INTERVENTIONS:
Drug: rosiglitazone

SUMMARY:
The purpose of this study is to gain safety and efficacy information in patients with type 2 diabetes, who have not previously taken any oral antidiabetic medications, and who have an HbA1c value of greater than or equal to 10%, despite diet and exercise.

ELIGIBILITY:
Inclusion criteria:

* Type 2 diabetes
* Drug-naive.
* Laboratory test result for HbA1c of greater than or equal to 10%.
* Written informed consent.

Exclusion criteria:

* Prior use of antidiabetic medications within 3 months of screening.
* Fluid retention (edema).
* Significant liver disease.
* Low red blood cells (anemia).
* Severe or unstable angina (chest pain).
* Congestive heart failure.
* Severe high blood pressure.
* Alcohol or drug abuse.
* Other inclusion or exclusion criteria to be determined by the physician and study sponsor.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142
Dates: Start 2002-05 (Actual); Primary Completion 2003-04-10 (Actual); Study Completion 2003-04-10 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline to Week 24.

SECONDARY OUTCOMES:
Change in FPG (fasting plasma glucose) from baseline to Week 24; characterize the effects of rosiglitazone on the albumin-creatinine ratio at Week 24.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Abstract: The Effects of Rosiglitazone in Poorly-Controlled, Drug-Naive Patients with Type 2 Diabetes Mellitus, KATHLEEN L. WYNE, ALEXANDER R. COBITZ, BRIAN R. WATERHOUSE, LEANNE J. STROW. Dallas, TX; King of Prussia, PA; Orlando, FL; USA. 64th Annual Scientific Sessions of the American Diabetes Association. 6/4/2004
- [Result] Wyne KL, Cobitz AR, Waterhouse BR, Strow LJ. The effects of rosiglitazone in poorly-controlled drug-naive patients with type 2 diabetes mellitus. Diabetes 2004;53(Suppl 2):A152. Poster 639 presented at ADA
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 49653/326 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 49653/326 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 49653/326 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 49653/326 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 49653/326 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 49653/326 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 49653/326 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register